CLINICAL TRIAL: NCT00904995
Title: Kinetics of 1, 3 Beta-d- Glucan Assay in Patients With Hematologic Malignancies Receiving Voriconazole Prophylaxis
Brief Title: Beta Glucan Assay in Patients Receiving Voriconazole Prophylaxis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0443
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Results first posted 2011-05-12 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Leukemia; Fungal Infection
Keywords: Leukemia; Cancer of the blood; Cancer of the bone marrow; Hematologic malignancy; Invasive fungal infection; Voriconazole; Vfend; antifungal prophylaxis
MeSH Terms: conditions — Leukemia; Mycoses; Hematologic Neoplasms; Invasive Fungal Infections | interventions — Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 - Oral (Experimental): Voriconazole Starting oral dose of 400 mg pills twice a day for first day, followed by 200 mg by mouth twice a day thereafter.
  Interventions: Drug: Voriconazole
- Group 2 - IV + Oral (Experimental): Voriconazole 6 mg/kg by vein (IV) first dose then 200 mg pills two times a day thereafter.
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Voriconazole — Starting dose of 400 mg by mouth twice a day for first day, followed by 200 mg by mouth twice a day thereafter.
  Other Names: Vfend
  Arms: Group 1 - Oral
Drug: Voriconazole — 6 mg/kg by vein for first dose, followed by 200 mg by mouth twice a day thereafter.
  Other Names: Vfend
  Arms: Group 2 - IV + Oral

SUMMARY:
Objectives:

To investigate the relationship between the administration of intravenous (IV) and oral voriconazole (vori) and the occurrence of false positive (1,3) beta-d- glucan (BG) relative to the standard assessment criteria used to diagnose invasive fungal infection in patients with hematologic malignancies.

DETAILED DESCRIPTION:
Chemotherapy can lower immune system function, which can cause fungal infections to occur more easily. These fungal infections are found by certain blood tests. One of these blood tests looks for a part of the fungal cell floating freely in the human blood.

When certain drugs are given to patients to prevent fungal infections, these blood tests may show that there is an infection when there actually is not one present. Some of these drugs are similar to the study drug voriconazole.

The Study Drug:

Voriconazole is designed to slow the growth of fungal cells, which may cause the fungal cells to die.

Screening Tests:

Signing this consent form does not mean that you will be able to take part in this study. You will have "screening tests" to help the doctor decide if you are eligible to take part in this study. The following tests and procedures will be performed:

* Your medical history will be recorded.
* You will have a complete physical exam.
* Blood (about 1 teaspoon) will be drawn for routine tests.
* If your doctor thinks it is needed, you will have a chest x-ray or computed tomography (CT) scan of the chest to check for pneumonia.

The study doctor will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in the study, you will not be enrolled. Other treatment options will be discussed with you.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to 1 of 2 study groups. Group 1 will consist of the first 10 patients enrolled on the study. Group 2 will consist of the next 10 patients enrolled on the study. If you are in Group 1, you will take only pills of study drug 2 times every day while you are on study. If you are in Group 2, you will receive the study drug through a needle in your vein 1 time when you begin the study and then take pills of study drug 2 times every day for the rest of the time you are on study.

Blood Draws for Fungal Infection Tests:

If you are in Group 1, blood (about 1 teaspoon each time) will be drawn for fungal infection tests at the following times:

* Before the first dose of study drug.
* 1, 2, 4, and 8 hours after the first dose of study drug.
* Before the third dose of study drug.
* 1, 2, 4, and 8 hours after the third dose of study drug.

If you are in Group 2, blood (about 1 teaspoon each time) will be drawn for fungal infection tests at the following times:

* Before the first dose of study drug.
* 1, 2, 4, and 8 hours after the first dose of study drug.
* 1, 2, and 4 hours after the second dose of study drug.

Length of Study:

You may continue taking the study drug for up to 35 days if you are receiving chemotherapy for the first time and up to 42 days if you have had chemotherapy before. Your doctor may decide that you should take the study drug for an even longer period of time or that you need to have another drug to prevent fungal infections. You will be taken off study if intolerable side effects occur or if you get a fungal infection.

Additional Information:

There are several drugs that should not be taken in combination with voriconazole. You should talk to the study doctor about any drugs you may be taking and about any drugs you may plan to start taking while on study. You should also avoid eating/drinking grapefruit/grapefruit products while you are on study, as they may interfere with the effects of the study drug.

This is an investigational study. Voriconazole is FDA approved and commercially available for the treatment of fungal infections.

Up to 20 patients who are found to be eligible after screening will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of hematologic malignancy with indication to receive antifungal prophylaxis.
2. Age >/= 18 years.
3. Patients must sign an informed consent.

Exclusion Criteria:

1. Patients with history of anaphylaxis attributed to azole compounds: voriconazole, itraconazole, fluconazole, posaconazole
2. Patients with clinical or other evidence that indicates that they have proven or probable invasive fungal infection prior to enrollment (European Organisation for Research and Treatment of Cancer (EORTC) criteria).
3. Patients with total bilirubin levels > 3 times the upper normal limits (i.e. > 3.0 mg/dl); or aspartate aminotransferase (AST or SGOT) or alanine aminotransferase (ALT or SGPT)> 5 times upper limit normal.
4. Patients receiving any medication that is contraindicated with the use of voriconazole. Voriconazole is contraindicated with the co-administration of the following drugs:sirolimus, terfenadine, astemizole, cisapride, pimozide, quinidine, ergot alkaloids, rifabutin, rifampin, high-dose ritonavir (400 mg Q12h), carbamazepine, long-acting barbiturates, efavirenz (with standard dose vfend and efavirenz), St. John's Wort.
5. Patients currently receiving voriconazole for antifungal prophylaxis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 4/2/09 to 8/19/09. All participants registered at The University of Texas M.D. Anderson Cancer Center.
Pre-assignment Details: Two of the twenty-three participants registered withdrew prior to their assignment to groups.
Period: Overall Study
Arm/Group | Group 1 - Oral | Group 2 - IV + Oral
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Oral | Group 2 - IV + Oral | Total
Number analyzed (Participants) | 10 | 11 | 21
Age Continuous [Median (Full Range); unit: years] | 52 [25 to 78] | 61 [20 to 76] | 56 [20 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Samples With BG Levels > 60pg/ml
Description: Rate calculated as number of participants with positive levels divided by total number of participants. beta-d-glucan (BG), a cell wall constituent of fungi, can be detected in serum as a marker of Invasive fungal infections (IFI).
  Blood samples were drawn on first 2 days of treatment at baseline (before the drug) and at 1, 2, 4, 8 hours after the first dose of the day. BG serum levels were measured using the Fungitell assay, using a cut off value of 60 pg/ml for positivity.
Time Frame: Up to 42 days
Population: Analysis was intent to treat with a total of 182 samples (mean 8.6 samples/participant) drawn from participants.
Measure: Number; unit: percent of blood samples
Units Other Than Participants: Blood samples
Arm/Group | Group 1 - Oral | Group 2 - IV + Oral
Number analyzed (Participants) | 10 | 11
Number analyzed (Blood samples) | 87 | 95
percent of blood samples
  Samples BG levels > 60pg/ml, First Test | 4 | 5
  Samples BG levels > 60pg/ml, Following Re-Test | 3 | 3

ADVERSE EVENTS:
Time Frame: 1 year 2 months
Arm/Group | Group 1 - Oral | Group 2 - IV + Oral
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes